CLINICAL TRIAL: NCT01802476
Title: A Phase 1, Single Dose, Fixed Sequence, 2-Period Cross-Over Absolute Oral Bioavailability Study In Healthy Volunteers Comparing Oral To Intravenous Administration Of PD-0332991
Brief Title: A Study Comparing the Plasma Drug Exposure of an Oral Dose of Palbociclib (PD-0332991) to an Intravenous Dose of Palbociclib (PD-0332991)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A5481015; QBR115052
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: PD-0332991; Absolute Bioavailability Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fixed Sequence Crossover Arm (Other): This study arm consists of a fixed sequence crossover where study subjects will receive Treatment A and following a washout of no less than 10 days will then receive Treatment B. The drug class is a CDK4/6 inhibitor.
  Interventions: Drug: Oral Drug Formulation of PD-0332991; Drug: Intravenous Formulation of PD-0332991

INTERVENTIONS:
Drug: Oral Drug Formulation of PD-0332991 — Treatment A consists of a single 125 mg oral dose of PD-0332991.
Drug: Intravenous Formulation of PD-0332991 — Treatment B consists of a 1000 mL intravenous infusion of 50 mg of PD-0332991 administered over 4 hours at a constant rate.

SUMMARY:
The purpose of this study is to determine approximately what percentage of an orally administered dose of PD-0332991 is absorbed from the gastrointestinal tract into the systemic circulation. This approximation is made by comparing the plasma pharmacokinetics of a 125 mg oral dose of PD-0332991 to the plasma pharmacokinetics of a 50 mg intravenous dose of PD-0332991 administered as a 4-hour infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female of non-childbearing potential between the ages of 18 and 55 years of age.
2. A body mass index (BMI) between 17.5 and 30.5 kg/m2, and a total body weight greater than 50kg (110 lbs)

Exclusion Criteria:

1. Any condition which could possibly affect drug absorption.
2. Pregnancy or actively nursing females, or females of childbearing potential.
3. A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Dose-Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0 to 144 hours
  Dose-Normalized AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8) divided by the administered dose. It is obtained from AUC (0 - t) plus AUC (t - 8).
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0 to 144 hours
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0 to 144 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Dose-Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0 to 144 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) divided by the administered dose.
Maximum Observed Plasma Concentration (Cmax) | 0 to 144 hours
Dose-Normalized Maximum Observed Plasma Concentration (Cmax) | 0 to 144 hours
  The maximum observed plasma concentration divided by the administered dose.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0 to 144 hours
Plasma Decay Half-Life (t1/2) | 0 to 144 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Systemic Clearance (CL) | 0 to 144 hours
  CL is a quantitative measure of the rate at which a drug substance is removed from the body following an intravenous dose.
Apparent Oral Clearance (CL/F) | 0 to 144 hours
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution after an Oral Dose (Vz/F) | 0 to 144 hours
Volume of Distribution at Steady State after an IV Infusion (Vss) | 0 to 144 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481015&StudyName=A%20Study%20Comparing%20the%20Plasma%20Drug%20Exposure%20of%20an%20Oral%20Dose%20of%20Palbociclib%20%28PD-0332991%29%20to%20an%20Intravenous%20Dose%20of%20Palbociclib%20%28PD